CLINICAL TRIAL: NCT00353158
Title: A Pilot Pediatric/Adult Study of Gene Expression Profiling and Clinical Characterization of Phototoxicity
Brief Title: A Pilot of Pediatric/Adult Study of Gene Expression Profiling and Clinical Characterization of Phototoxicity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 060198; 06-AR-0198; NCT00411008 (obsolete NCT alias)
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-26

CONDITIONS: Healthy Volunteers; Fungal Infections; Bacterial Infections
Keywords: Phototesting; UVR/UVA; Sunburn; Doxycycline; Voriconazole
MeSH Terms: conditions — Mycoses; Bacterial Infections; Sunburn | interventions — Doxycycline; Voriconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A (Active Comparator): Subjects currently on or previously on chronic voriconazole or subjects who are scheduled to begin voriconazole
  Interventions: Drug: Voriconazole
- B (Experimental): 100mg twice daily for 3 days. Two hours after the last dose of doxycycline is taken in the clinic, on-medication phototesting with ssUVR, UVA, and visible light will be performed.
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — 100mg twice daily for 3 days. Two hours after the last dose of doxycycline is taken in the clinic, on-medication phototesting with ssUVR, UVA, and visible light will be performed.
  Arms: B
Drug: Voriconazole — After taking voriconazole for (Bullet)7 days to achieve a steady state of voriconazole for subjects, on-medication phototesting with ssUVR, UVA, and visible light will be performed.
  Arms: A

SUMMARY:
This study will examine the phototoxicity, a reaction to light that is like exaggerated sunburn, which occurs in people who take medications such as voriconazole, a medication used to fight fungus. Sunscreens might protect the skin from the reaction. Although phototoxicity from voriconazole is not completely understood, it may be related to how that medication is metabolized in the liver by enzymes called cytochrome P450 enzymes-and mainly by one known as 2C19. A way to evaluate phototoxicity is through microarrays, which measure how much each gene is expressed in cells from tissues such as skin.

Patients ages 8 and older who are scheduled to begin taking or who currently take voriconazole may be eligible for this study. Also, patients ages 18 to 45 in good health who have skin tone known as Type 2, which usually burns and tans only slightly following sun exposure, may be eligible. All patients will visit the Dermatology Clinic. They will complete two questionnaires, on medical history and medications, as well as the skin response to sunlight, and donate about 3 teaspoons of blood. Patients who are scheduled to take voriconazole will visit the clinic four times, that is, two visits 2 consecutive days before beginning the medication and two visits on 2 consecutive days after taking it for at least 7 days. Each visit will take 1 to 2 hours. Patients about to take voriconazole will have a blood test and undergo a physical exam of the skin test site, on the buttocks. Researchers will take photographs of the specific site and do tests to measure skin reaction to ultraviolet (UV) light. UV light will be shined on 15 small areas of the skin, each 1 x 1 centimeters. After 24 hours, any redness that occurs on the skin will be checked. Afterward, patients will begin taking voriconazole according to directions by the researchers. At 10 or more days later, patients will visit the clinic. Sunscreen will be applied and 1 hour later after administration of voriconazole, a blood sample will be drawn to check the level of medication. Then UV light will be shined on 23 areas of skin 1 x 1 centimeters. More photographs will be taken of test sites to record changes in skin redness. On the next day, the skin response will be evaluated. Participants in the control group will be asked to avoid UV radiation by wearing hats and clothing, and using sunscreen. They will be given the doxycycline, an antibiotic, and undergo procedures with UV light shined on small areas of the skin, on the buttocks. Control participants will have 7 study days, with visits lasting from 1 to 3 hours and probably not exceeding 8 hours. They will have two shave biopsies on Study Day 2 and on Study Day 7 to determine how the skin has responded to UV light exposures.

...

DETAILED DESCRIPTION:
Background:

* Phototoxicity is a sunburn-like response associated with certain medications and is a phenomenon which is not completely understood. Although clinically similar to a typical sunburn reaction, the gene expression changes in phototoxic skin reactions may differ from those in typical sunburn.
* Doxycycline is a relatively well-tolerated and known phototoxic antimicrobial which can be used in healthy volunteers to increase susceptibility to phototoxicity.
* Characterizing potential risk factors to phototoxicity secondary to voriconazole, a broad-spectrum antifungal agent associated with potentially treatment-limiting phototoxicity, may allow identification of subjects at risk for the adverse reaction via pharmacogenetic evaluation and medical record review.
* Subjects at risk of phototoxicity may benefit from application of effective sunscreens.

Objectives:

* To determine the global gene expression profiles in skin exhibiting phototoxic reactions in healthy volunteers treated with doxycycline, and compare expression profiles in skin exposed to ultraviolet (UV) radiation occurring in the absence of doxycycline.
* To investigate the effects of the doxycycline alone in the skin of phototoxic and non-phototoxic healthy volunteers.
* To characterize voriconazole-related phototoxicity reactions in subjects with the use of phototesting and to determine if these subjects may receive reasonable phototoxic protection from the use of sunblock.

Eligibility:

* I & II) Healthy volunteers with skin phototype II.
* III) Subjects scheduled to begin voriconazole therapy.
* IV) Subjects on chronic voriconazole with or without a history of phototoxicity reaction.
* Previously treated healthy volunteers (I & II) who were evaluated to be either phototoxic

OR non-phototoxic.

Design:

* I) For the Screening visit arm, forty healthy volunteers will undergo screening with pertinent skin exam and blood work to evaluate ANA/ENA and liver function profile.
* II) For the Study visit arm, eligible healthy volunteers will undergo phototesting and will have skin biopsies prior to initiating a 3-day course of oral doxycycline 100 mg twice daily.
* After the last dose of doxycycline, healthy volunteers will undergo on-treatment MED testing.
* In those demonstrating phototoxicity, skin biopsies will be performed and submitted for processing for microarray analysis.
* III) Thirty-five subjects scheduled to begin voriconazole will undergo CYP450 genotyping and baseline phototesting prior to initiation of voriconazole.
* Adult subjects will be invited to undergo optional skin biopsies pre-drug and on-drug.
* Repeat phototesting will be performed in subjects after at least 7 days of voriconazole to determine if voriconazole predisposes to phototoxicity.
* Subjects with voriconazole phototoxicity will be invited to undergo sunscreen testing.
* IV) Seventy subjects with prior clinical history of voriconazole phototoxicity as well as known voriconazole phototoxicity non-reactors will undergo CYP450 genotyping and potential phototesting.
* To investigate the effects of the doxycycline alone in the skin of healthy volunteers previously categorized as phototoxic and non-phototoxic

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects who are scheduled to begin voriconazole

1. Subjects with any skin phototype who are scheduled to begin voriconazole therapy.
2. Availability of unexposed skin for testing. Test sites for ssUVR, UVA, and visible light exposures should be devoid of sunburn, suntan, scars, active dermal lesions, prior radiotherapy exposure, and uneven skin tones. The presence of nevi will be acceptable if in the physician's judgment they will not interfere with the study results. (Excess hair is acceptable if clipped or shaved.)
3. Ages >= 8 years old.
4. Ability to participate fully and comply with the procedures of the protocol in the opinion of the investigator.
5. Ability of subjects or guardians to understand and sign the consent form. Children must give assent for participation in addition to parental consent.

OR

Subjects currently on or previously on chronic voriconazole

1. Subjects with any skin phototype who have received or are currently receiving chronic voriconazole therapy.
2. Ages >= 8 years old.
3. Ability to participate fully and comply with the procedures of the protocol in the opinion of the investigator.
4. Ability of subjects or guardians to understand and sign the consent form. Children must give assent for participation in addition to parental consent.

OR

Healthy volunteers

I) Screening visit arm.

1. Healthy adults aged 18-45 year old of skin phototype II (age and skin phototype limits selected to simulate subjects evaluated in protocol 04-C-0120).
2. No history of allergy to tetracyclines.
3. No systemic medications, herbal supplements or vitamins that are known to be associated with abnormal light response or effect on cytochrome P450 enzymes taken concurrently or within 7 days or 7 half-lives (whichever is longer) of phototesting.
4. No history of liver disease or hepatitis.
5. Willing to undergo screening dermatologic examination and bloodwork.
6. Ability to understand and sign the consent form.

II) Study visit arm

1. Anti-nuclear antibodies (ANA) <3 EU; Negative extractable nuclear antigen (ENA); and negative history of idiopathic abnormal response to sunlight, such as polymorphic light eruption or solar urticaria. Prior remote history of phototoxicity reactions acceptable.
2. Availability of unexposed skin for testing. Test sites for ssUVR, UVA, and visible light exposures should be devoid of sunburn, suntan, scars, active dermal lesions, prior radiotherapy exposure, and uneven skin tones. The presence of nevi will be acceptable if in the physician's judgment they will not interfere with the study results. (Excess hair is acceptable if clipped or shaved.)
3. Liver function profile must be within limits of normal.
4. Ability to participate fully and comply with the procedures of the protocol in the opinion of the investigator.

EXCLUSION CRITERIA:

Subjects who are scheduled to begin voriconazole

1. Does not meet the inclusion criteria.
2. Extensive skin disease and no testable skin area available.
3. History of allergic reactions to lidocaine for the adults who will undergo the modified shave biopsy.
4. History of idiopathic abnormal response to sunlight, such as polymorphic light eruption or solar urticaria. Prior remote history of phototoxicity reaction allowed.
5. Unable to comply with the requirements of the protocol.
6. Any confounding past or present medical illness that in the judgment of the investigators would pose added risk for study participants (i.e. subjects with history of graft-versus-host disease; subjects on concurrent chemotherapy or completed chemotherapy within the preceding two weeks with known photoexacerbating agents such as alkylating agents, doxorubicin, methotrexate, or cisplatin; or subjects with previous radiotherapy to the intended sites for phototesting).
7. Pregnancy.
8. History of keloid formation in the adults who will undergo the modified shave biopsy.

OR

Subjects currently on or previously on chronic voriconazole

1. Does not meet the inclusion criteria.
2. Unable to comply with the requirements of the protocol.
3. Any confounding past or present medical illness that in the judgment of the investigators would pose added risk for study participants.

OR

Healthy volunteers

I) Screening visit arm.

1. Does not meet the Screening visit arm inclusion criteria.
2. History of allergic reactions to lidocaine.
3. Any confounding past or present medical illness that in the judgment of the investigators would pose added risk for study participants (i.e. subjects with history of graft-versus-host disease; subjects on concurrent chemotherapy with known photoexacerbating agents such as alkylating agents, doxorubicin, methotrexate, or cisplatin; or subjects with previous radiotherapy to the intended sites for phototesting).
4. Pregnancy.
5. History of keloid formation.

II) Study visit arm

1. Does not meet the Study visit arm inclusion criteria.
2. Extensive skin disease and no testable skin area available.
3. Anti-nuclear antibodies (ANA) >= 3 EU or positive extractable nuclear antigen (ENA); prior history of idiopathic abnormal response to sunlight, such as polymorphic light eruption or solar urticaria. Prior remote history of phototoxicity reaction allowed.
4. Unable to comply with the requirements of the protocol.

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-05-25 (Actual); Primary Completion 2011-09-20 (Actual); Study Completion 2011-09-20 (Actual)

PRIMARY OUTCOMES:
Global gene expression profiles | After treatment with voriconazole/doxycycline
  fully evaluable microarray sets of doxycycline-associated phototoxic reactions

CONTACTS AND LOCATIONS:
Overall Officials: Heidi H Kong, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-AR-0198.html